CLINICAL TRIAL: NCT06219824
Title: Clinical and Radiographic Evaluation of Bioceramic Putty Mineral Trioxide Aggregate Versus Mineral Trioxide Aggregate in Pulpotomy of Immature Permanent Molars: A Randomized Clinical Trial
Brief Title: Clinical and Radiographic Evaluation of Bioceramic Putty MTA Versus MTA in Pulpotomy of Immature Permanent Molars
Acronym: MTA
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Marwa Abd El-Naby Hussien, Assistant lecturer of Pediatric Dentistry, Faculty of Dentistry, October University for Modern Sciences and Arts, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14422022599195
Record Dates: First submitted 2024-01-01; First posted 2024-01-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Pulpotomy; Deep Caries
Keywords: Immature permanent molars,; young permenent molars; pulpotomy; vital pulp therapy; deep caries; Putty MTA; bioceramic MTA

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- control Group (Active Comparator): pulpotomy treatment for the young permanent teeth will be done using conventional powder and liquid Mineral Trioxide Aggregate followed by Glassionomer restoration and stainless steel crown
  Interventions: Drug: Conventional MTA
- Experimental (Experimental): pulpotomy treatment for the young permanent teeth will be done using premixed ready for use bioceramic MTA followed by Glassionomer restoration and stainless steel crown
  Interventions: Drug: premixed Bio-ceramic MTA

INTERVENTIONS:
Drug: premixed Bio-ceramic MTA — pulpotomy treatment will be done and the premixed bioceramic MTA will be applied in the pulp chamber
  Other Names: well Root MTA
  Arms: Experimental
Drug: Conventional MTA — pulpotomy treatment will be done and powder and liquid MTA will be mixed and applied in the pulp chamber
  Other Names: Pro-root MTA
  Arms: control Group

SUMMARY:
The present study aims to evaluate the clinical and radiographic success of bioceramics putty MTA versus MTA in the pulpotomy of immature permanent molars

The main question it aims to answer is:

Will the biocermaics putty MTA have higher clinical and radiographic success rates than MTA in pulpotomy of immature permanent molars?

DETAILED DESCRIPTION:
limited clinical trials have reported the clinical and radiographic outcomes after pulpotomy with premixed putty bioceramic MTA and conventional MTA in young permanent molars.

MTA has various drawbacks, such as difficulty in handling, long setting time, discoloration of the tooth, and its form as a powder/liquid which raise the responsibility for major material waste. To conquer these issues, bioceramic materials have been developed premixed putty bioceramic MTA is a ready-to-use material for immediate placement with zero waste, saving cost and chair time. Thus, the present study aims to evaluate bioceramic putty MTA's clinical and radiographic success versus MTA in pulpotomy of immature permanent molars.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged from 6-8 years of both sexes have immature permanent molars
* with deep carious lesions indicated for pulpotomy.
* Restorable young permanent molars with no clinical symptoms of irreversible pulpitis.
* Permanent molars without any clinical sign of pulp necrosis including swelling, fistula, pain on percussion, and pathologic tooth mobility.
* Permanent molars without any adverse radiographic findings including thickening of the periodontal ligament space, radiolucency at the interradicular or periapical regions
* permanent molars without internal and external root resorption, or calcification in pulp tissue.

Exclusion Criteria:

* Medically compromised patients who have systemic disease.
* Uncooperative patients who refuse treatment.
* Permanent molars that were previously restored.

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome | 24hrs, 1 week
  Immediate Postoperative pain [ Time Frame: one week) post operative pain by Verbal analogue scale.It is a 10 cm long horizontal line with points labeled from 0 to 10 where (0) indicates no pain, (1-3) mild pain, (4-6) moderate pain, and (7-10) severe pain.

SECONDARY OUTCOMES:
Secondary outcome | 6,12 month
  The increase in root length, The root lengthening will be assessed in Mm through Digora software

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No